CLINICAL TRIAL: NCT04490161
Title: Prevention of Cerebral Vasospasm Following Aneurysmal Subarachnoid Hemorrhage Through Treatment With Intravenous Autologous Cerebrospinal Fluid - a Pilot Trial.
Brief Title: Prevention of Vasospasm in SAH Through CSF Treatment
Acronym: PREVAIL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1193/2018
Record Dates: First submitted 2020-04-30; First posted 2020-07-28 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-07

CONDITIONS: Subarachnoid Hemorrhage; Subarachnoid Hemorrhage, Aneurysmal; Vasospasm, Cerebral; Aneurysmal Subarachnoid Hemorrhage
Keywords: EVD; Aneurysm; SAH; Subarachnoid hemorrhage; cerebral vasospasm; cerebrospinal fluid
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Subjects will receive reinstallation of CSF intravenously.
  Interventions: Other: intravenous reinstallation of cerebrospinal fluid
- Observational (No Intervention): Subjects will not receive study intervention; CSF will be sampled and analyzed in comparison to the Interventional arm,

INTERVENTIONS:
Other: intravenous reinstallation of cerebrospinal fluid — 10ml of CSF will be taken under sterile conditions from the external ventricular drain and immediately administered intravenously.
  Arms: Interventional

SUMMARY:
The pathophysiological mechanisms of aneurysmal subarachnoid haemorrhage (aSAH) involve early brain injury (EBI) and delayed cerebral ischemia (DCI).

Several mechanisms contribute to EBI pathogenesis, including cell death, inflammatory response, oxidative stress, excitotoxicity, microcirculatory dysfunction, microthrombosis and cortical spreading depolarization. All are suggested to be linked due to common pathogenic pathways and direct interaction.

Despite advances in research of diagnostics and treatment strategies, brain injury remains the major cause of death and disability in SAH patients. There is no sufficient treatment of SAH and its devastating consequences known so far. Developing and improving diagnostic methods to monitor SAH patients and to evaluate efficacy of treatment strategies are essential in SAH research. These include neuroimaging, biomarkers, and other parameters such as invasive multimodal neuromonitoring and intraoperative electrophysiological monitoring.

Cerebral vasospasm (CV) - mostly responsible for DCI - can be depicted on angiograms. Altogether, tremendous efforts have been taken to conquer the occurrence and sustainability of CV. The mortality of patients suffering aSAH rises up to 50% if the patients' condition is critical (Hunt&Hess (HH) Grade 5, WFNS Grade 5, modified Fisher Grade 4).

Reports of beneficial outcome in patients with pre-existing CSF shunting have been published. The hypothesis of early CSF reapplication to the bloodstream, in order to prevent CV seems to be positively approved by the mentioned reports. Nevertheless, no data could be found on the mechanisms of action in this phenomenon.

To confirm the presence of interaction of the mechanisms of EBI and evaluate the application of cerebrospinal fluid (CSF), a pilot clinical trial was planned. Due to the lack of validated animal models for aSAH it is necessary to perform the trial first-in-human. A pilot (proof of concept) trial - is done through inclusion of 10 patients with severe aSAH (≥HH4). According to clinical guidelines, these patients receive external ventricular drainages in order to drain CSF and lower intracranial pressure. An interim analysis of data will be performed after inclusion and treatment of 5 patients. Blood-/CSF-sampling for further analysis will be collected before, during and after treatment according to the study protocol.

DETAILED DESCRIPTION:
Aneurysmal subarachnoid haemorrhage (aSAH) is associated with high morbidity and mortality with an incidence of 5-9 per 100,000 population. The incidence of aSAH peaks amongst those of 40-60 years1; aSAH carries a high overall mortality rate of up to 67%2 with only around half of the survivors able to live independently. Given the age-related incidence 3 and high morbidity and mortality, SAH has a high burden on society . Conventionally following SAH, treatment is directed to securing the aneurysm to prevent further re-bleed. In addition to the primary brain injury due to the rupture of the aneurysm the occurrence of cerebral vasospasm (VS) with narrowing of the brain supplying arteries potentially lading to brain ischemia is as well - known and serious complication following aSAH. The development of VS is thought to be caused by various factors. Interestingly, this is not an instant phenomenon occurring right after the hemorrhagic event. VS develops rather in a time dependent fashion with a peak incidence around 7-10 days following from acute event.

From angiographic studies, it is known that up to 70% of all patients with a aSAH will develop VS and in about 40% of these it will result in clinical deterioration and in 10-15% in permanent delayed ischemic neurologic deficits (DIND) leading to an increased morbidity 4, 5 and mortality

. Based on the fact that VS develops with a time delay, this is thought to provide a "therapeutic window" allowing to initiate measures for its prevention. However, in spite of intensive experimental and clinical research the investigators still do not have any effective treatment for the prevention of VS in patients with aSAH. Many concepts have been elaborated in the past, mostly based o sound pharmacologic considerations such as calcium antagonists (Nimodipin), antioxidants (Tirilazad) and endothelin antagonists (Clazosentan). In clinical trials, however, none of these drugs have shown a therapeutic effect on VS and most of them have been abandoned since then. The only exception is the use of oral Nimodipin, which is still used showing a marginal effect 6-8.

In contrast to all previous studies, which were based on the use of specific drugs, the present hypothesis is different. It is based on the assumption that the brain is a "privileged" organ, where the in- and outflow is regulated by discrete barrier mechanisms (e.g. blood-brain- barrier). In the event of aSAH - factors that are thought to play an important role in the development of VS are released into the CSF. However, it is not clear whether these factors will enter the systemic circulation. This is further supported by the clinical observation that in many patients with aSAH, acute disturbances of CSF circulation can be seen, often resulting in hydrocephalus. This in return can be treated by CSF flow diversion with the use of external ventricular drainage, which is a routine procedure in the management of aSAH patients.

Based on the assumption that those factors responsible for the development of VS are contained in the CSF, but do not enter the systemic circulation, it then might make sense to use the externally drained CSF for intravenous re-administration and thereby activating a systemic response mechanism with in turn could prevent the development of VS.

The potential therapeutic benefits outweigh any potential risks for patients with aSAH.

The proposed clinical study involves autologous CSF without any changes made to the liquid. The CSF will be taken from the external ventricular drain (EVD) under sterile environment and reinfused intravenously.

An interval of approximately 21 days will permit a timely review and evaluation of interim safety (after 5 patients) and tolerability data collected The potential benefit to patients is significant with reduced delayed cerebral infarction (DCI), improved cognition and cerebral function. As such, studies in patients with aSAH are warranted, with a view to establishing the optimal dose, safety and exploratory efficacy profiles.

This is a pilot trial involving higher grade (see inclusion criteria) aSAH patients.

The human brain is protected and enjoying privileged immune status. The blood-brain- barrier (BBB) leads to consequent isolation of brain tissue from humoral immunity. The brain is experiencing several major changes during rupture of a cerebral aneurysm. First, the intracranial pressure increases immediately, caused by the actual bleeding. Second, the extravasation of blood disrupts the BBB and several immunogenic molecules travel through the spontaneous rupture into the CSF. Additionally, microscopic particles of the vessel wall are present in the CSF as a consequence of the wall rupture. Usually, these potentially spasmogenic fractions are never encountered by the brain and the external surface of its vessels. Interestingly, the perioperative collection of blood in subarachnoid spaces does not induce vasospasm.

The investigators hypothesized that the reported steps were crucial for the formation of cerebral vasospasm.

This study will be conducted in compliance with the protocol and according to Good Clinical Practice and applicable regulatory standards. No deviation from the protocol will be implemented without the prior review and approval by the relevant ethics and regulatory authorities, except where it may be necessary to eliminate an immediate hazard to a research subject. In such case, the deviation will be reported to the relevant ethics and regulatory authorities as soon as possible.

Ten patients with an angiographically confirmed aSAH, who in addition are in need of early external ventricular drainage (routine procedure), irrespective of the clinical grade on admission and in whom definite treatment (clip ligation or interventional treatment) is achievable within 72 hours following aSAH.

Following aneurysm clip ligation, the predetermined amount of CSF (10ml) will be obtained under sterile conditions directly from the external ventricular drain and administered in a peripheral vein. To reduce the possibility of contamination, the application of CSF will be done immediately. In case of extensive intraventricular hemorrhage, causing the aspiration of clotted blood while obtaining CSF, the patient needs to be excluded from the trial.

A number of patients will have an EVD placed for clinical reasons. These patients would regularly have CSF sampling ranging from daily to twice weekly.

In this study, approximately 2 ml CSF will be taken and stored for translational study purposes (starting on day of EVD fitting) until day 21 or until the EVD is removed as per standard of care.

ELIGIBILITY:
Inclusion Criteria:

Age: >18, <90

* SAH HH 3 - 5
* Cerebral saccular Aneurysm
* Digital subtraction angiography prior to aneurysm repair
* Aneurysm repair within 72h
* Modified Fisher Grade 3+4
* Presence of aneurysm needing treatment (clipping or coiling)
* Treatment within 24 hours of symptom onset
* External ventricular drain (clinical need)

Exclusion Criteria:

* Non-aneurysmal SAH

  * SAH HH<3
  * Extensive intraventricular haemorrhage (unable to obtain CSF without massive aspiration of clotted blood)
  * Contraindication for digital subtraction angiography
  * Aneurysm repair >72h after rupture
  * Signs of radiographic vasospasm upon diagnosis
  * Presence of systemic or CSF infection
  * Contraindication for oral Nimodipin
  * Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe radiographic vasospasm | 8 (+/- 1) day post SAH
  measured upon digital subtraction angiography

SECONDARY OUTCOMES:
Infectious complications | 7 days
  presence of infections complications according to the study intervention (intravenous administration)
Incidence of vasospasm-related morbidity / mortality | within 21 days post-aneurysm securing
  Defined by on of the following: DIND (confirmed by mGCS); cerebral infarction upon CT scan (day 14), need for anti-vasospasm therapy within 14 day post securing

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Rooij NK, Linn FH, van der Plas JA, Algra A, Rinkel GJ. Incidence of subarachnoid haemorrhage: a systematic review with emphasis on region, age, gender and time trends. J Neurol Neurosurg Psychiatry. 2007 Dec;78(12):1365-72. doi: 10.1136/jnnp.2007.117655. Epub 2007 Apr 30. PMID 17470467
- [Background] Nieuwkamp DJ, Setz LE, Algra A, Linn FH, de Rooij NK, Rinkel GJ. Changes in case fatality of aneurysmal subarachnoid haemorrhage over time, according to age, sex, and region: a meta-analysis. Lancet Neurol. 2009 Jul;8(7):635-42. doi: 10.1016/S1474-4422(09)70126-7. Epub 2009 Jun 6. PMID 19501022
- [Background] Kreiter KT, Copeland D, Bernardini GL, Bates JE, Peery S, Claassen J, Du YE, Stern Y, Connolly ES, Mayer SA. Predictors of cognitive dysfunction after subarachnoid hemorrhage. Stroke. 2002 Jan;33(1):200-8. doi: 10.1161/hs0102.101080. PMID 11779911
- [Background] Connolly ES Jr, Rabinstein AA, Carhuapoma JR, Derdeyn CP, Dion J, Higashida RT, Hoh BL, Kirkness CJ, Naidech AM, Ogilvy CS, Patel AB, Thompson BG, Vespa P; American Heart Association Stroke Council; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular Nursing; Council on Cardiovascular Surgery and Anesthesia; Council on Clinical Cardiology. Guidelines for the management of aneurysmal subarachnoid hemorrhage: a guideline for healthcare professionals from the American Heart Association/american Stroke Association. Stroke. 2012 Jun;43(6):1711-37. doi: 10.1161/STR.0b013e3182587839. Epub 2012 May 3. PMID 22556195
- [Background] Langham J, Reeves BC, Lindsay KW, van der Meulen JH, Kirkpatrick PJ, Gholkar AR, Molyneux AJ, Shaw DM, Copley L, Browne JP; Steering Group for National Study of Subarachnoid Haemorrhage. Variation in outcome after subarachnoid hemorrhage: a study of neurosurgical units in UK and Ireland. Stroke. 2009 Jan;40(1):111-8. doi: 10.1161/STROKEAHA.108.517805. Epub 2008 Nov 13. PMID 19008474
- [Background] Pickard JD, Murray GD, Illingworth R, Shaw MD, Teasdale GM, Foy PM, Humphrey PR, Lang DA, Nelson R, Richards P, et al. Effect of oral nimodipine on cerebral infarction and outcome after subarachnoid haemorrhage: British aneurysm nimodipine trial. BMJ. 1989 Mar 11;298(6674):636-42. doi: 10.1136/bmj.298.6674.636. PMID 2496789
- [Background] Dorhout Mees SM, Rinkel GJ, Feigin VL, Algra A, van den Bergh WM, Vermeulen M, van Gijn J. Calcium antagonists for aneurysmal subarachnoid haemorrhage. Cochrane Database Syst Rev. 2007 Jul 18;2007(3):CD000277. doi: 10.1002/14651858.CD000277.pub3. PMID 17636626
- [Background] Vergouwen MD; Participants in the International Multi-Disciplinary Consensus Conference on the Critical Care Management of Subarachnoid Hemorrhage. Vasospasm versus delayed cerebral ischemia as an outcome event in clinical trials and observational studies. Neurocrit Care. 2011 Sep;15(2):308-11. doi: 10.1007/s12028-011-9586-8. PMID 21748502
- [Background] Vergouwen MD, Vermeulen M, van Gijn J, Rinkel GJ, Wijdicks EF, Muizelaar JP, Mendelow AD, Juvela S, Yonas H, Terbrugge KG, Macdonald RL, Diringer MN, Broderick JP, Dreier JP, Roos YB. Definition of delayed cerebral ischemia after aneurysmal subarachnoid hemorrhage as an outcome event in clinical trials and observational studies: proposal of a multidisciplinary research group. Stroke. 2010 Oct;41(10):2391-5. doi: 10.1161/STROKEAHA.110.589275. Epub 2010 Aug 26. PMID 20798370